CLINICAL TRIAL: NCT04744116
Title: A Randomized Controlled Pilot Study of Two Doses of Cord Blood Tissue-Derived Mesenchymal Stromal Cells Combined With Ruxolitinib Versus Ruxolitinib Alone for Therapy of Steroid-Refractory Acute Graft Versus Host Disease
Brief Title: Addition of Cord Blood Tissue-Derived Mesenchymal Stromal Cells to Ruxolitinib for the Treatment of Steroid-Refractory Acute Graft Versus Host Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1122; NCI-2020-13889 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1122 (Other: M D Anderson Cancer Center); P01CA148600 (NIH)
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Steroid Refractory Graft Versus Host Disease
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Cell- and Tissue-Based Therapy; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (ruxolitinib) (Active Comparator): Patients receive ruxolitinib PO BID for at least 3 days and may consider tapering after 6 months of therapy if response occurs and therapeutic corticosteroid doses have been discontinued.
  Interventions: Drug: Ruxolitinib
- Arm 2 (ruxolitinib, lower dose ds-MSCs) (Experimental): Patients receive ruxolitinib PO BID as in Arm 1. Patients also receive lower dose of cb-MSCs IV for up to 60 minutes twice weekly (at least 3 days apart) over 4 consecutive weeks for 8 total doses.
  Interventions: Other: Cellular Therapy; Drug: Ruxolitinib
- Arm 3 (ruxolitinib, higher dose ds-MSCs) (Experimental): Patients receive ruxolitinib PO BID as in Arm 1. Patients also receive higher dose of cb-MSCs IV for up to 60 minutes twice weekly (at least 3 days apart) over 4 consecutive weeks for 8 total doses.
  Interventions: Other: Cellular Therapy; Drug: Ruxolitinib

INTERVENTIONS:
Other: Cellular Therapy — Given ds-MSCs IV
  Other Names: Cell Therapy
  Arms: Arm 2 (ruxolitinib, lower dose ds-MSCs); Arm 3 (ruxolitinib, higher dose ds-MSCs)
Drug: Ruxolitinib — Given PO
  Other Names: INCB-18424; INCB18424; Jakafi; Oral JAK Inhibitor INCB18424

SUMMARY:
This early phase I trial is to find out the effect of adding cord blood tissue-derived mesenchymal stromal cells (cb-MSCs) to ruxolitinib in treating patients with acute graft versus host disease that does not respond to steroid therapy (steroid-refractory). Ruxolitinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. cb-MSCs are a type of tissue helper cell that can be removed from donated umbilical cord blood tissue and grown into many different cell types that can be used to treat cancer and other disease, such as graft versus host disease. This trial aims to learn if adding cb-MSCs to ruxolitinib may help control steroid-refractory acute graft versus host disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate between-arm differences (Arm 3 versus [vs] Arm 1, and Arm 2 vs Arm 1) for each of the 28-day co-primary outcome probabilities.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM 1: Patients receive ruxolitinib orally (PO) twice daily (BID) for at least 3 days and may consider tapering after 6 months of therapy if response occurs and therapeutic corticosteroid doses have been discontinued.

ARM 2: Patients receive ruxolitinib PO BID as in Arm 1. Patients also receive lower dose of cb-MSCs intravenously (IV) for up to 60 minutes twice weekly (at least 3 days apart) over 4 consecutive weeks for 8 total doses.

ARM 3: Patients receive ruxolitinib PO BID as in Arm 1. Patients also receive higher dose of cb-MSCs IV for up to 60 minutes twice weekly (at least 3 days apart) over 4 consecutive weeks for 8 total doses.

After completion of study treatment, patients are followed up on day 28 and then for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Participants between the ages of 12 years and 80 years (inclusive).
2. Steroid refractory grades II-IV acute GVHD of the Lower GI tract or Liver (including those developing these manifestations after previous acute GVHD of skin) secondary to allogeneic HCT or donor lymphocyte infusion. (Grading, see Appendix I) GVHD with: No improvement after treatment with methylprednisolone at ≥ 2.0 mg/kg/day or equivalent for minimum 7 days, or progressive symptoms after minimum 3 days, or a flare in acute GVHD while on systemic steroids. Participants must have had a biopsy that suggests GVHD; a repeat biopsy to enroll on the study is not necessary.
3. Karnofsky/Lansky Performance score of at least 30 at the time of study entry.
4. Participants who are women of childbearing potential, must be non-pregnant, not breast-feeding, and use adequate contraception. Male patients must use adequate contraception
5. Participants (or legal representative where appropriate) must be capable of providing written informed consent, and assent if indicated.

Exclusion Criteria:

1. De novo chronic GVHD
2. Isolated acute GVHD of skin
3. Secondary systemic therapy for acute GVHD ruxolitinib greater than 96 hours before initiation of therapy.
4. Primary treatment with agents other than alpha-1 antitrypsin (AAT) glucocorticoids and ruxolitinib.
5. Participants with uncontrolled infections will be excluded. Infections are considered controlled if appropriate therapy has been instituted and, at the time of enrollment, no signs of progression are present. Progression of infection is defined as hemodynamic instability attributable to sepsis, new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
6. Adult and pediatric patients with cognitive impairments and/or any serious unstable pre-existing medical condition or psychiatric disorder that can interfere with safety or with obtaining informed consent or compliance with study procedures.
7. Participants with significant supplemental oxygen requirement defined as >6 L oxygen by nasal cannula.
8. Participants with known allergy to bovine or porcine products.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Death from any cause | Within 28 days from the start of active study treatment
Response | At day 28 from start of therapy on study
  Will compare the patient's 28-day graft versus host disease (GVHD) status to the patient's baseline GVHD status when steroid refractory acute GVHD was diagnosed.
Incidence of adverse events | Within 28 days from the start of active study treatment

SECONDARY OUTCOMES:
Graft versus host disease status | At days 7, 14, 21 and 28 post treatment
  Will assess complete response (CR), very good partial response (VGPR), partial response (PR), stable disease (SD), and progressive disease (PD).
Proportion of response | At days 7, 14, 21 and 28 post treatment
  Will assess proportion of patients with CR, PR, VGPR, and no-response (NR). The event NR is defined as stable disease, mixed response, disease progression, OR initiation of additional systemic (second-line) GVHD therapies.
Time to complete response | Up to 6 months
  Will be estimated by the method of Kaplan and Meier.
Time to very good partial response | Up to 6 months
  Will be estimated by the method of Kaplan and Meier.
Time to partial response | Up to 6 months
  Will be estimated by the method of Kaplan and Meier.
Incidence of complete response for each organ | Up to 6 months
Incidence of very good partial response for each organ | Up to 6 months
Incidence of partial response for each organ | Up to 6 months
Durability of organ response | Up to 6 months
Cumulative incidence of non-relapse mortality (NRM) | At 6 months post treatment
Cumulative incidence of relapse/progression of the primary disease | At 6 months
Overall survival | From enrollment to death from any cause, assessed at 6 months
Disease-free survival | From enrollment to death from any cause or relapse/progression of the primary disease, assessed at 6 months
Graft versus host disease-free survival | At 6 months
  Patients alive, free of active acute or chronic GVHD, and without other systemic agents (or escalation of steroids to >= 2.5 mg/kg/day of prednisone [or methylprednisolone equivalent of 2 mg/kg/day]) added for treatment of GVHD will be considered successes for this endpoint
Incidence of chronic graft versus host disease | At 6 months after first mesenchymal stromal cells (MSC) infusion
  Chronic GVHD is defined per National Institutes of Health Consensus Criteria. Diagnosis of chronic GVHD of any severity (mild, moderate, or severe) is considered an event for this endpoint. Organ involvement and maximum severity will also be described at six months.
Incidence of systemic infections | 28 days after last study drug
  The incidence of grade 2 to 3 systemic infections occurring from study treatment until 28 days after last study drug will be described using standard Common Terminology Criteria for Adverse Events (CTCAE) criteria. Infections will be recorded by site of disease, date of onset, and severity.
Incidence of toxicities | Up to 28 days after completing last MSC infusion study drug
  The incidence of grade 3-5 treatment-emergent adverse events (per CTCAE version 5.0) that occur through 28 days after completing last MSC infusion study drug will be described.
Incidence of any grade cytokine release | Up to 28 days after completing last MSC infusion study drug
Incidence of any infusional toxicity | Within 24 hours of each cord blood-MSC infusion

OTHER OUTCOMES:
Cytokine biomarker analysis (optional) | Up to 6 months
  Will use cytokine biomarker assays to predict response to therapy.
Fecal samples analysis (optional) | Up to 6 months
  Will use fecal samples to assess microbiome and potential predictor for response to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Partow Kebriaei, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org